CLINICAL TRIAL: NCT00768014
Title: fMRI Measurements on the Effect of Transcutaneous Electrical Nerve Stimulation (TENS) on Acupuncture Points Verses Spontaneous Normal Vaginal Delivery to Relief of Labor Pain
Brief Title: fMRI Measurements on Pain Relief Methods in First Stage Labor Pain
Acronym: TENS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: AS Chao, MD, Chang Gung Memorial Hospital
Other Study IDs: 97-1707B; YY Wai; JJ Wang; ZH Wang
Record Dates: First submitted 2008-10-05; First posted 2008-10-07 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Labor Pain; Pain Relief; Magnetic Resonance Imaging
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Healthy term pregnant women in labor without any pain relief
- 2: Healthy term pregnant women received TENS
- 3: Healthy term pregnant women received epidural anesthesia

SUMMARY:
The purposes of this study is to integrate the objective tests into the subjective test, visual analog score (VAS), for evaluation and further understanding of relieving labor pain by TENS application on acupuncture points in the first stage of labor.

DETAILED DESCRIPTION:
Our published paper "Pain relief by applying transcutaneous electrical nerve stimulation (TENS) on acupuncture points during the first stage of labor: a randomized double-blind placebo-controlled trial. (Pain 2007; 127:214-20 )" about the double-blind randomized placebo-controlled study, sponsored by NSC 91-2314-B-182A-162-grant in 2002, showed that TENS application on acupuncture points resulted in significantly better pain relief than placebo by visual analogue scale (VAS) score in the first stage of labor. Two hurdles that hampered physicians to evaluate the possible therapies in the management of obstetric pain. Firstly, there is no objective test for pain. Secondly, lack of controlled trials for different analgesic methods of pain treatment (interventional, psychological, physical therapy).

Transcutaneous electrical nerve stimulation (TENS) is one of the non-pharmacological means of pain relief for labor and delivery. We aimed to investigate the efficacy and safety of TENS on specific acupuncture points for reducing pain in the first stage of labor. In this double-blind, placebo-controlled trial, we randomly assigned healthy full-term parturients in active phase of first-stage labor to either TENS on 4 acupuncture points (Hegu [Li 4] and Sanyinjiao [Sp 6].

Visual analogue scale (VAS) will be used as an adjunct objective assessment of pain relief efficacy by having a scale with a range from 1 to 10, where 1 represented no pain and 10 the most painful. Participants will be asked by study personnel to estimate how painful during the last contractions before the application of TENS, 30 minutes and 60 minutes after TENS application. VAS will be recorded at each application (first, second application, and so forth) as described till the end of first stage. Within 24 hours after delivery, the women will be asked to fill in a questionnaire regarding the satisfaction of pain relief using TENS during labor. Augmentation of labor will be administered to achieve three uterine contractions in 10 minutes in the first stage according to the protocol of induction of labor. Continuous external electronic fetal heart rate monitoring and tocodynamometry are used for fetal surveillance. Polygraph recording of maternal heart rate, transcutaneous oxygen tension, respiratory rate will be used for evaluate the changes. Details of the effect of analgesia in participants switching to it, the progression of cervical dilation and the length of first stage after the application of TENS are recorded. The request for epidural anesthesia or other form of analgesia will be available upon request. Adverse events such as discomfort of movement restriction, skin allergy, or electrical accident were recorded if any. Decision of performing operative delivery was made only according to maternal and fetal indications. fMRI A scan will be collected in between 30-60 minutes after the application TENS. Subjects will be asked to lie supine on the scanner bed and motion artifact will be excluded. MR imaging parameters: Functional scans using 3.0-Tesla Siemens Allegra MRI System equipped for echo-planar imaging. Blood oxygenation level-dependent (BOLD) functional imaging will be carried out using a gradient echo T2-weighted pulse sequence. At least 38 sagittal slices, 3 mm thick with 0.6-mm gap will be performed in each scan. Image collection was preceded by four dummy scans to allow for equilibration of the MRI signal. A3D MPRAGE T1-weighted high-resolution structure dataset was collected before functional imaging to facilitate Talairach transformation and visualization.

ELIGIBILITY:
Inclusion Criteria:

* an initial wish to deliver without epidural analgesia
* primigravida
* planned vaginal childbirth without obstetrical or non-obstetrical complications
* fetal vertex presentation
* term pregnancy (>37 weeks of gestation)
* age between 20 and 40 years
* no experience in acupuncture or TENS for other reasons
* no previous poor obstetrical outcome (either maternal or fetal). For those subjects willing to have fMRI: This study will be carried out only on right-handed Chinese women under accompany by a family member.

Exclusion Criteria:

* psychiatric and neurologic disorders,
* candidate for vaginal birth after cesarean (VBAC); and
* head trauma with loss of conscious,
* major medical illness e.g., pacemaker parturient.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-07 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: An-Shine Chao, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- AS Chao, Guishan, Tao-Yuan, Taiwan